CLINICAL TRIAL: NCT06447441
Title: Clinical Outcomes Of Mega-dosage Supplementations Of Cholecalciferol In Critically Ill Patients With Sepsis
Acronym: MDC-S
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Collaborators: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Chin-Ming Chen, M.D., Professor, Chimei Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMMC11302007
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Critically Ill; Sepsis; Mortality Rate; Critical Care
Keywords: Vitamin D; Cholecalciferol; Sepsis
MeSH Terms: conditions — Critical Illness; Sepsis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Enteral supplementation of placebo in 3 days
  Interventions: Other: Placebo
- Vitamin D3 group (Experimental): Enteral supplementation of 1,728,000 IU vitamin D3 in 3 days
  Interventions: Other: Cholecalciferol

INTERVENTIONS:
Other: Placebo — Enteral supplementation of placebo in 3 consecutive days within 96 hours after ICU admission.
  Arms: Placebo
Other: Cholecalciferol — Enteral supplementation of 576,000IU/day vitamin D3 in 3 consecutive days within 96 hours after ICU admission
  Other Names: vitamin D3
  Arms: Vitamin D3 group

SUMMARY:
Non-COVID-19 sepsis (Sepsis) has always been one of the common diseases in critically ill patients. The main treatment strategy is to kill pathogens and mitigate hyperinflammation. One study demonstrated that the supplementation with 576,000 IU cholecalciferol (vitamin D3) as a single dose in critically ill adults in the medical intensive care units (MICUs) can improve clinical outcomes, including acute physiology and chronic health evaluation II score (APACHE II), sequential organ failure assessment score (SOFA), and C-reactive protein (CRP).

It is a three-year, multi-center, prospective, parallel, double-blind, randomized controlled clinical trial for 240 eligible subjects, with administrations of vitamin D3 576,000 IU or placebo every 24 hours for 3 days (72 hours) within 96 hours after intensive care unit (ICU) admission.

ELIGIBILITY:
Inclusion Criteria:

1. Medical subject ≥ 18 years old and diagnosed with sepsis
2. Transferred to the intensive care unit within 24 hours after being diagnosed with sepsis
3. Admitted to the ICU with 40 > APACHE II score ≥ 15.
4. The intensivist anticipates that the subject will stay in the ICU ≥ 7 days.

Exclusion Criteria:

1. Diseases that affect serum levels of 25(OH)D and calcium, including thyroidectomy, parathyroid disease, rickets, or severe cirrhosis [Child C]
2. Received large doses of vitamin D3 in the past four weeks (> 2000 IU per day or ≥ 10,000 IU in a single dose)
3. Admitted to the ICU with diagnosis of COVID-19
4. AIDS subjects taking immunosuppressants
5. Organ transplant
6. Active cancer
7. Tuberculosis, sarcoidosis, or kidney stones in the past one year
8. Weight < 45 kg or > 90 kg
9. Had been admitted to ICU in the past three months
10. Subject and family members who do not speak the native language
11. Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day Mortality | Up to 30 days after intervention
  Duration from the day of intervention to subjects died

SECONDARY OUTCOMES:
ICU Length of Stay of Survivors | Up to 30 days after intervention
  Duration from the day of intervention to ICU discharge
iPTH concentration | 12 hours pre-intervention, Day5-6 post-intervention, Day15-16 pre-intervention, Day 29-30 post-intervention (or the day ICU discharge)
calcifediol concentration ( 25(OH)D ) | 12 hours pre-intervention, Day5-6 post-intervention, Day15-16 pre-intervention, Day 29-30 post-intervention (or the day ICU discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Chin Ming Chen, Principal Investigator — Chimei Medical Center

IPD SHARING:
Plan to Share IPD: No